CLINICAL TRIAL: NCT07280702
Title: Deucravacitinib-TNF Combination Therapy for Difficult-to-Control Psoriatic Disease
Acronym: COMBo
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Merola, Professor & Chair-Dermatology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2025-0977
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Psoriatic Arthritis (PsA)
Keywords: Psoriatic Arthritis; PsA; Deucravacitinib; TNF
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- established standard of care anti-TNF plus deucravacitinib (Experimental): Deucravacitinib will be administered in tablet form. Anti-TNF will be administered by injection.
  Interventions: Drug: Deucravacitinib
- established standard of care anti-TNF plus placebo (Placebo Comparator): Placebo will be administered in tablet form. Anti-TNF will be administered by injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Drug will be administered in tablet form.
  Arms: established standard of care anti-TNF plus deucravacitinib
Drug: Placebo — Drug will be administered in tablet form.
  Arms: established standard of care anti-TNF plus placebo

SUMMARY:
The purpose of this research study is to determine the effectiveness of adding deucravacitinib to the participant's current Psoriatic Arthritis (PsA) treatment to see if it improves their symptoms and quality of life.

This study is exploring a new treatment approach that may help improve control of psoriatic disease by targeting different parts of the disease process. By combining therapies that work together, the goal is to offer better symptom relief with fewer or more manageable side effects than some current treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 with confirmed psoriatic arthritis based on CASPAR criteria.

  * Ability to provide informed consent and comply with study procedures.
  * Patients with plaque psoriasis BSA>3% OR PsA with [SJC>2 AND TJC >3] despite stable background anti-TNF therapy for at least 6 months, with or without csDMARDs (i.e MTX, leflunomide, sulfasalazine, hydroxychloroquine).
  * Concurrent use of 1 csDMARD, and/or NSAID, and/or oral glucocorticoid is permitted but not required during the study. If such treatment was administered, then participants must meet the following requirements:

    * If on csDMARD (methotrexate [MTX], sulfasalazine [SSZ], leflunomide [LEF], hydroxychloroquine [HCQ]), the participant must have been on it for at least 12 weeks and be on a stable dose for at least 28 days prior to Day 1.

      * If on MTX, the route of administration and dose must be stable and the dose must be ≤ 25 mg/week.
      * If on SSZ, the dose must be ≤ 3 g/day.
      * If on HCQ, the dose must be ≤ 400 mg/day.
      * If on LEF, the dose must be ≤ 20 mg/day. Note: If currently not on MTX, SSZ, or HCQ, the participant must not have received it for at least 28 days prior to Day 1. If currently not on LEF, the participant must not have received it for at least 12 weeks prior to Day 1.
    * If on an NSAID, the participant must be on a stable dose for at least 14 days prior to Day 1.
    * Stable background use of prednisone 15 mg daily or equivalent is permitted. If on oral glucocorticoids, the participant must be on a stable dose of ≤ 15 mg/day prednisone equivalent for at least 28 days prior to Day 1.
    * Note: If currently not on oral glucocorticoids, the participant must not have received oral glucocorticoids within 28 days prior to Day 1

Exclusion Criteria:

* History of failure of more than two anti-TNF therapies, prior history of failure of TYK2 and JAK inhibitors.

  * History of prior allergic reaction or intolerance to deucravacitinib.
  * History of primary failure of anti-IL17, anti-IL23 is excluded. Note that prior exposure to these agents is allowed for reasons other than primary failure, eg intolerance, insurance / access issues, etc).

    * Systemic agents other than anti-TNF or csDMARD (ie. MTX, leflunomide, sulfasalazine, hydroxychloroquine) must have ceased > 6 months prior to baseline.
    * Doses or glucocorticoids >15mg daily prednisone or equivalent.
  * Severe cardiovascular, hepatic, or renal impairment.
  * History or evidence of outpatient active infection and/or febrile illness within 14 days prior to Day 1.
  * History of serious bacterial, fungal, or viral infection requiring hospitalization or parenteral antimicrobial treatment (eg, antibiotics antiviral, antifungal, or antiparasitic agents) within 60 days prior to Day 1.
  * Receipt of any therapy for chronic infection (eg, pneumocystis, herpes zoster, cytomegalovirus, invasive bacterial or fungal infections, or atypical mycobacteria) at screening.
  * Recent herpes zoster or herpes simplex infection or history of serious herpes zoster or herpes simplex infection defined as:
  * a) Herpes zoster or herpes simplex lesions within 30 days prior to randomization, OR
  * b) History of serious herpes zoster or serious herpes simplex infection, which includes, but it is not limited to, any episode of disseminated herpes simplex, multi- dermatomal herpes zoster, herpes encephalitis, ophthalmologic herpes, and/or recurrent herpes zoster (recurrent herpes zoster is defined as more than 2 episodes in the last 2 years).
  * Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status (eg, history of opportunistic infections [eg, Pneumocystis jirovecii pneumonia, histoplasmosis, or coccidioidomycosis], history of splenectomy, primary immunodeficiency).
  * Receipt of any live vaccine within 60 days prior to Day 1 or plans to receive a live vaccine during the study or within 60 days after completing study treatment.
  * Evidence of, or positive testing for, hepatitis B virus or hepatitis C virus at screening.
  * Positive testing for human immunodeficiency virus 1 or 2 by antibody testing at screening.
  * History of active TB prior to the screening visit, signs or symptoms of active TB at screening, positive QuantiFERON®-TB Gold (or equivalent) test result or 2 successive indeterminate QuantiFERON®-TB Gold (or equivalent) test results at screening.
  * History of chronic or recurrent infectious disease.
  * History of VTE, MACE, active solid malignancy or history of malignancy <5 years, any hematologic malignancy; history of multiple serious infections requiring hospitalization in the past 5 years, history of opportunistic infection, any condition which in the opinion of the investigator would pose a safety risk or inability to assess key endpoints in the study.
  * History of fibromyalgia/central sensitization, or other joint disease which in the opinion of the investigator would make musculoskeletal disease activity assessment challenging in the context of this study.
  * History of other inflammatory dermatosis which in the opinion of the investigator would make skin disease activity assessment challenging in the context of this study (eg atopic, contact dermatitis, etc).
  * Exclude use of topicals except for mild to mid-potency topical steroids for use only in cosmetically sensitive areas such as the face.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a novel composite endpoint of BSA </= 1 AND SJC </= 1) OR (BSA </= 1 AND TJC </= 1) at 24 weeks | 24 weeks
  Proportion of patients achieving a novel composite endpoint of BSA </= 1 AND SJC </= 1) OR (BSA </= 1 AND TJC </= 1) at 24 weeks

SECONDARY OUTCOMES:
Safety and tolerability, measured through adverse event reporting at baseline and weeks 5, 12, 24, and 48. | baseline and weeks 5, 12, 24, and 48
  Safety and tolerability, measured through adverse event reporting at baseline and weeks 5, 12, 24, and 48.
Proportion of patients achieving Minimal Disease Activity (5/7 criteria) at weeks 24 and 48 | weeks 24 and 48
  Reaching Minimal Disease Activity involves achieving 5 of 7 criteria. The 7 criteria include less than or equal to 1 tender joint count, patient global assessment of disease activity via Visual Analog Scale of less than or equal to 20, less than or equal to 1 swollen joint count, tender entheseal points of less than or equal to 1, Psoriatic Area and Severity Index of less than or equal to 1 OR Body Surface Area of less than or equal to 3 %, patient pain via Visual Analog Scale of less than or equal to 15, and Health Assessment Questionnaire - Disability Index of less than or equal to 0.5. The Minimal Disease Activity assessment will be done at weeks 24 and 48.
Proportion of patients achieving Very Low Disease Activity (7/7 criteria) at weeks 24 and 48 | weeks 24 and 48
  Very Low Disease Activity involves achieving 7 of 7 criteria. The 7 criteria include less than or equal to 1 tender joint count, patient global assessment of disease activity via Visual Analog Scale of less than or equal to 20, less than or equal to 1 swollen joint count, tender entheseal points of less than or equal to 1, Psoriatic Area and Severity Index of less than or equal to 1 OR Body Surface Area of less than or equal to 3 %, patient pain via Visual Analog Scale of less than or equal to 15, and Health Assessment Questionnaire - Disability Index of less than or equal to 0.5. The Very Low Disease Activity assessment will be done at weeks 24 and 48.
Proportion of patients achieving Minimal Disease Activity - Skin (MDA with skin domain met) at weeks 24 and 48 | weeks 24 and 48
  Minimal Disease Activity - Skin is determined by a Psoriatic Area and Severity Index of less than or equal to 1 OR Body Surface Area of less than or equal to 3 %. The Minimal Disease Activity - Skin assessment will be done at weeks 24 and 48.
Percentage achieving Psoriatic Area and Severity Index 75/90/100, PASI < 1 BL at weeks 12, 24 and 48 | baseline and weeks 12, 24 and 48
  75%, 90% and 100% improvement in Psoriatic Area and Severity Index of less than 1 at baseline. This assessment will be done at weeks 12, 24 and 48.
Percentage achieving BSA < 1% (NPF definition) BL at weeks 12, 24 and 48 | baseline and weeks 12, 24 and 48
  Percentage achieving BSA < 1% (NPF definition) BL at weeks 12, 24 and 48
Resolution of Spondyloarthritis Research Consortium of Canada at baseline and at weeks 24 and 48 | baseline and weeks 24 and 48
  Resolution of Spondyloarthritis Research Consortium of Canada at baseline and at weeks 24 and 48
Resolution of Leeds Enthesitis Index at baseline and at weeks 24 and 48 | baseline and weeks 24 and 48
  Resolution of Leeds Enthesitis Index at baseline and at weeks 24 and 48
Change from baseline Health Assessment Questionnaire - Disability Index at weeks 24 and 48 | baseline and weeks 24 and 48
  Change from baseline Health Assessment Questionnaire - Disability Index at weeks 24 and 48
Change from baseline Pruritis Numeric Rating Scale at weeks 12, 24 and 48 | baseline and weeks 12, 24 and 48
  Change from baseline Pruritis Numeric Rating Scale at weeks 12, 24 and 48
Change from baseline Joint pain Visual Analog Scale at weeks 12, 24 and 48 | baseline and weeks 12, 24 and 48
  Change from baseline Joint pain Visual Analog Scale at weeks 12, 24 and 48
Change from baseline patient global assessment of arthritis at weeks 12, 24 and 48 | baseline and weeks 12, 24 and 48
  Change from baseline patient global assessment of arthritis at weeks 12, 24 and 48
Change from baseline Dermatology Life Quality Index at weeks 12, 24 and 48 | baseline and weeks 12, 24 and 48
  Change from baseline Dermatology Life Quality Index at weeks 12, 24 and 48
Change from baseline Psoriatic Arthritis Impact of Disease 12-item Questionnaire and proportion achieving Patient Acceptable Symptom State cutoff at weeks 12, 24 and 48 | baseline and weeks 12, 24 and 48
  Change from baseline Psoriatic Arthritis Impact of Disease 12-item Questionnaire and proportion achieving Patient Acceptable Symptom State cutoff at weeks 12, 24 and 48

OTHER OUTCOMES:
Leed's enthesitis (resolution) BL at weeks 24 and 48 | baseline and weeks 24 and 48
  Leed's enthesitis (resolution) BL at weeks 24 and 48
Widespread pain index at baseline and at weeks 24 and 48 | baseline and weeks 24 and 48
  Widespread pain index at baseline and at weeks 24 and 48
International Dermatology Outcome Measure Musculoskeletal Questionnaire instrument (instrument validation) at baseline and at weeks 12, 24 and 48 | baseline and weeks 12, 24 and 48
  International Dermatology Outcome Measure Musculoskeletal Questionnaire instrument (instrument validation) at baseline and at weeks 12, 24 and 48
Cardiometabolic biomarker evaluation at baseline, week 24 and week 48 | baseline, week 24 and week 48
  Cardiometabolic biomarker evaluation includes tests for lipids, glycoprotein acetylation, fasting glucose, insulin levels, hemoglobin A1c, C-Reactive Protein, homeostatic model assessment for insulin resistance. These tests will be done at baseline, week 24 and week 48
Symptom Severity Scale (used for post-hoc stratification analyses) at baseline and at weeks 24 and 48 | baseline and at weeks 24 and 48
  Symptom Severity Scale (used for post-hoc stratification analyses) at baseline and at weeks 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Merola, MD MMSc, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided